CLINICAL TRIAL: NCT04064359
Title: A Phase I, Open-label, Dose Finding Study to Assess the Safety, Tolerability, PK, and Preliminary Efficacy of OBT076, a CD205-directed ADC, in Recurrent and/or Metastatic CD205+ Solid Tumors
Brief Title: Safety and Preliminary Efficacy of OBT076 in Recurrent/Metastatic CD205+ Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford BioTherapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OBT076-001
Record Dates: First submitted 2019-08-16; First posted 2019-08-21 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OBT076 Dose Escalation and Expansion (Experimental): OBT076 administered intravenously (IV) every 3 weeks in escalating dose cohorts during Part A and OBT076 administered at or below the MTD in the Part B expansion cohort. In Part C sequential administration of OBT076 administered at the recommended phase 2 dose (RP2D) followed by Balstilmab. Part D will evaluate the safety, tolerability, preliminary efficacy of OBT-076 in combination with Balstilmab. Part E will evaluate the safety, tolerability and preliminary efficacy of OBT076 as a triple combination regimen with balstilimab and gemcitabine in patients with metastatic NSCLC (Cohort E1) or locally-advanced/metastatic urothelial cancer Cohort E2)
  Interventions: Drug: OBT076, a CD205-directed antibody-drug conjugate

INTERVENTIONS:
Drug: OBT076, a CD205-directed antibody-drug conjugate — Intravenous (IV) infusion of OBT076 every 3 weeks.
  Other Names: MEN1309

SUMMARY:
The purpose of this study is to evaluate OBT076, which is a drug that combines an antibody with an anti-cancer drug. This class of drugs are called Antibody-Drug Conjugates (ADC). Antibodies are normally produced in the human body by the immune system to fight infections but can be designed to target cancer cells and deliver an anti-cancer drug. OBT076 is composed of an antibody that targets the CD205 protein on cancer cells and delivers an anti-cancer drug which can kill them. OBT076 is an "Investigational Drug", which means that it is still being studied and has not yet been approved by the US Food and Drug Administration (FDA), the European Medicines Agency (EMA) or any other regulatory authorities to be prescribed by doctors for the treatment of metastatic or recurrent solid tumors. The use of OBT076 in this study is investigational.

This is a Phase I research study designed to look at several dose levels of the study drug to find the highest dose level that is safe and well-tolerated (does not cause unacceptable side effects), and to examine the effects of the study drug in a small group of research participants. The study will also look at the effectiveness of OBT076 as an anti-cancer therapy. Once the optimal dose is determined and safety is assessed, additional research participants will be treated at the optimal dose level to further evaluate safety and effectiveness.

DETAILED DESCRIPTION:
Study OBT076-001 is an open-label, Phase I, dose escalation and expansion clinical study of OBT076 in CD205+ve recurrent and/or metastatic solid tumors that are refractory to standard treatments, or for which a standard therapy is not available or not suitable or is no longer effective. The study will consist of four parts:

* Part A: Dose escalation
* Part B: OBT076 single agent expansion
* Part C: Sequential administration of OBT076 and balstilimab
* Part D: Combination therapy with concurrent administration of OBT076 and balstilimab• Part E: Triple combination therapy with concurrent administration of OBT076, balstilimab and gemcitabine in two cohorts of patients with metastatic NSCLC or locally-advanced/metastatic urothelial cancer.

Parts A, B, C, D will and E consist mainly of 3 periods: Screening, Treatment and Follow-up periods. The treatment period with OBT076 consists of 21 days cycles. Approximately 200 patients will be enrolled across Parts A to E.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 years of age (at the time of signing the ICF) with non-curative recurrent and/or metastatic solid tumors for which a standard therapy is not available or is no longer effective.
2. Subject has histologically and/or cytologically confirmed solid tumors.
3. Subject with Breast cancer:

   1. Subject with hormone-receptor positive (as per local laboratory) recurrent locally advanced or metastatic breast cancer, regardless of HER2 status, must have received at least two prior lines of endocrine therapy in the adjuvant or metastatic setting, either as monotherapy or in combination with targeted therapy
   2. Subject with recurrent locally advanced or metastatic non-curative HER2 negative breast cancer (based on most recently analyzed biopsy), HER2 status is defined as per ASCO-CAP guidelines as negative, if in situ hybridization test or IHC status is 0, 1+, or 2+.
   3. Subject with triple negative breast cancer are eligible after at least one prior line of cytotoxic chemotherapy in the metastatic setting.
   4. Subject with prior adjuvant or neoadjuvant chemotherapy allowed.
4. Subject has received a maximum of two prior lines of cytotoxic chemotherapy in the metastatic setting. Subject who received three up to five prior lines of cytotoxic chemotherapy in the metastatic setting are eligible, if the last administration of cytotoxic chemotherapy was at least 12 weeks prior to Cycle 1 Day 1
5. Subject has tumor that is positive for CD205 antigen by IHC staining
6. Subject has an ECOG performance status of 0-1.
7. Subject has radiological documented measurable disease (i.e., at least 1 measurable lesion as per RECIST Version 1.1).
8. Subject has adequate organ function
9. Subject has adequate bone marrow function
10. Subject understands and voluntarily signs an ICD prior to any study-related assessments/procedures are conducted.
11. Subject is able to adhere to the study visit schedule and other protocol requirements.
12. Subject who is a female of childbearing potential (defined as a sexually mature women, has not undergone hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal for at least 12 consecutive months and is using any adequate form of birth control must:

    1. Have a negative pregnancy test within 1 week before first dose of study drug.
    2. Use highly effective method(s) of birth control consistently and correctly during the study and for at least 4 months after the last dose of study drug.
    3. Agree to not donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for at least 4 months after the last dose of study.
    4. Agree to no plan to breastfeed and no plan to become pregnant during the study and for at least 4 months after the last dose of study drug.
13. Subject who is a sexually active male must agree to use a condom, not to donate sperm and have no plans to father a child during the study and for at least 4 months after the last dose of study drug.

Exclusion Criteria:

1. Subject has received any chemotherapy within 28 days prior to Cycle 1 Day 1.
2. Subject has received any other systemic anticancer therapy within 28 days or 5 half-lives of Cycle 1 Day 1.
3. Subject has symptomatic visceral crisis requiring chemotherapy per Investigator judgment for non TNBC.
4. Subject with colorectal cancer and pancreatic cancer are not eligible for the study.
5. Subject with peritoneal involvement, i.e., peritoneal carcinomatosis, are not eligible for the study.
6. Subject has not recovered from the acute toxic effects (CTCAE grade ≤ 1) of prior anticancer therapy, radiation, or major surgery/significant trauma (except alopecia or other toxicities not considered a safety risk for the subject at the Investigator's discretion).
7. Subject has had major surgery within 14 days prior to starting study treatment or has not recovered from major side effects.
8. Subject has had radiotherapy ≤ 4 weeks prior to starting study drug.
9. Subject has a history of, or current symptomatic brain metastasis.
10. Subject has any other malignancy within 5 years prior to randomization
11. Subject has a known or suspected hypersensitivity or other contraindication to any excipients used in the manufacture of OBT076.
12. Subject has significant medical condition, laboratory abnormality, or psychiatric illness that would, in the Investigator's judgment, contraindicate patient participation in the study (e.g., history of thromboembolic event, cardiac dysfunction, chronic pancreatitis, chronic active hepatitis)
13. Subject has severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine <7 days before Cycle 1 Day 1
14. Subject has any condition that confounds the ability to interpret data from the study.
15. Subject is lactating or breastfeeding.
16. Subject has a past medical history of or ongoing clinically relevant interstitial lung disease, drug-induced pneumonitis or severe/very severe COPD.
17. Subject has active or chronic corneal disorder or Sjogren's syndrome.
18. Subject has any ongoing skin disorders not controlled by specific treatment.
19. Subject has significant active cardiac disease within the previous 6 months including unstable angina or angina requiring surgical or medical intervention, significant cardiac arrhythmia, or NYHA class 3 or 4 congestive heart failure, or patients with QTc interval >470ms at screening.
20. Subject has a known history or current diagnosis of HIV infection, unless on triple antiviral treatment with undetectable viral load.
21. Subject who is female of childbearing potential
22. Subject who is unable or unwilling to take folic acid or vitamin B12 supplementation.
23. Subject with a history of allogeneic organ transplant.
24. Subject with grade 3 or 4 immune-related adverse reactions during any prior line of checkpoint inhibitor containing therapy. Patients with immune-related thyroiditis controlled with substitution, or prior asymptomatic lipase increases are eligible for the study.
25. Subject with active autoimmune disease or history of autoimmune disease that required systemic treatment within 3 years of the start of study treatment.

Additional inclusion criteria specific for Part E:

1. Patients with stage IV NSCLC or stage III/stage IV urothelial cancer who have progressed on standard treatments or for whom a standard therapy is not available, standard therapy is no longer effective, or who have no satisfactory treatment options.

Additional exclusion criteria for Part E:

1. The presence of any contraindication to gemcitabine as per applicable Summary of Product Characteristics/label.
2. Patients with a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalent) within the 14 days prior to the first dose of study treatment or another immunosuppressive medication within the 30 days prior to the first dose of study treatment. Inhaled or topical steroids, and adrenal replacement steroid doses )\ mg daily prednisone equivalent) are permitted in the absence of active autoimmune disease.
3. Patients with urothelial cancer and any history or current CNS metastasis.
4. Patients who were hospitalized during screening for infectious complications or required IV antibiotics in the 14 days prior to Cycle 1 Day 1.
5. Patients who presented in the 14 days prior to or on Cycle 1 Day 1 with one or more of the following:

   * ANC of <1.5 x 109 cells/L
   * Platelets of < 100 x 109 cells/L
   * Hemoglobin of < 9 g/dL
6. Patients who received G-CSF in the 14 days prior to Cycle 1 Day 1
7. Patients who had febrile neutropenia during the previous line of therapy or during the last line of therapy containing cytotoxic chemotherapy.
8. Patients who are primary refractory to anti-PD-(L)1 directed therapy.
9. Patients with NSCLC and more than 2 prior lines of systemic anti-cancer therapy in the locally-advanced/metastatic disease setting; and who received more than one prior line of cytotoxic chemotherapy in the locally-advanced/metastatic setting.
10. Patients with urothelial cancer who received more than 3 prior lines of systemic anti cancer therapy in locally-advanced/metastatic disease setting. Prior neoadjuvant or adjuvanttherapy is not counted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) as assessed by NCI CTCAE (Version 5) | 1 year
  Assess incidence of all AEs by NCI CTCAE (Version 5) grades 1-5
Percentage of subjects with dose-limiting toxicities (DLTs) as assessed by NCI CTCAE (Version 5) | 1 year
  DLTs defined by NCI CTCAE (Version 5) grades 3-4, with exceptions for duration

SECONDARY OUTCOMES:
Clinical Benefit Ratio (CBR) | 2 years
  RECIST, Version 1.1
Overall Response Rate (ORR) | 2 years
  RECIST, Version 1.1
Duration of Response (DoR) | 2 years
  Kaplan-Meier methodology
Progression Free Survival (PFS) | 2 years
  Kaplan-Meier methodology
Overall Survival (OS) | 2 years
  Kaplan-Meier methodology
Area under the Plasma Concentration versus Time Curve (AUC) of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076
Maximum Plasma Concentration [Cmax] of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076
Time Taken to Reach the Maximum Plasma Concentration [Tmax] of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076
Half-Life [T1/2] of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076
Clearance (CL) of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076
Volume of Distribution (Vd) of OBT076 | 1 year
  Statistics including number of subjects (N), mean, standard deviation, CV%, geometric mean, geometric CV%, median, minimum, and maximum will be provided for OBT076

OTHER OUTCOMES:
Quantification of Serum Protein | 2 years
  Enzyme-linked Immunosorbant Assay (ELISA)
Quantification of Peripheral Blood CD205+ Cells | 2 years
  Flow Cytometry
Quantification of Immune Cells (ICs) in Tumor Microenvironment (TME) | 2 years
  Immunohistochemistry

CONTACTS AND LOCATIONS:
Locations (27):
- United States (10):
  - Mayo Clinic, Phoenix, Arizona
  - Cedars-Sinai, Los Angeles, California
  - UCLA, Santa Monica, California
  - Moffitt Cancer Center, Tampa, Florida
  - The State University of Iowa, Iowa City, Iowa
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Quantum Santa Fe, Santa Fe, New Mexico
  - Columbia University Medical Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - AZ Groeninge, Kortrijk
- France (7):
  - Institut Paoli Calmettes, Marseille
  - GHP Saint-Joseph, Paris
  - Hopital Saint Antoine, Paris
  - Hopital Saint Louis, Paris
  - Centre Eugène Marquis, Rennes
  - ICANS - Institut de cancérologie Strasbourg, Strasbourg
  - Institut Gustave Roussy - IGR, Villejuif
- Greece (5):
  - University General Hospital Attikon, Chaïdári, Athens
  - Metropolitan Hospital, Athens
  - Sotiria General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - EuroMedica, Thessaloniki
- Spain (3):
  - START Barcelona HM Nou Delfos, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - University Hospital Marqués de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: No